CLINICAL TRIAL: NCT03411928
Title: Modified Endotracheal Balloon Dilator to Improve Oxygenation During Airway Procedures in Children With Tracheal Stenosis
Brief Title: Endotracheal Dilator to Improve Oxygenation
Acronym: EDITION2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Red Cross War Memorial Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Ross Hofmeyr, Associate Professor, Dept Anaesthesia & Perioperative Medicine, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCT_ENT_Anaes_201801
Record Dates: First submitted 2018-01-09; First posted 2018-01-26 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Tracheal Stenosis; Airway Disease; Pediatric Respiratory Diseases
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Intervention Model Description: Prospective interventional study
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracheolator (Experimental): Tracheal dilatation using the study device as per the protocol.
  Interventions: Device: Tracheolator

INTERVENTIONS:
Device: Tracheolator — 'Tracheolator' non-occlusive tracheal dilation balloon manufactured by Disa Life Sciences, Cape Town, South Africa.

SUMMARY:
The purpose of the study is to prospectively assess the use of a modified tracheal balloon dilator in children (<13 years old) with subglottic or tracheal stenosis. The hypothesis is that the device will effectively dilate the stenotic segment, whilst maintaining oxygenation (if applicable). The primary aim is to measure the stenosis prior to, and after dilatation; using diameter and the modified Myer-Cotton grading system. Secondary aims include assessment of stenosis at six-week follow-up and monitoring arterial oxygenation nadir (using peripheral plethysmography) during the procedure.

DETAILED DESCRIPTION:
This study is a prospective, single arm, observational study of patients at Red Cross War Memorial Children's Hospital receiving treatment for laryngotracheal stenosis using a modified tracheal dilatation balloon. The tracheal balloon dilatation procedure is clinically well-established and is standard practice in the study institution. In this study, a modified, improved tracheal balloon will be used to treat patients. Data to be collected during the procedure include measurement of the stenotic segment prior to and after dilatation, using both the modified Myer-Cotton grading system and sizing the stenosis using endotracheal tubes diameter, documenting the site of the stenosis (distance from vocal cords), periprocedural oxygen saturation nadir (using plethysmography) and heart rate. All other procedures will be as per routine care. Each procedure will be monitored by a senior anaesthetist who is not a member of the research team. Their role will be to ensure the safety of the patient.

The tracheal balloon dilatation device consists of a catheter tube which has an inflation port at its proximal end and a balloon at its distal end. The balloon is provided in a narrow, folded condition to allow entering and traversing the stenotic portion of the airway. As with all tracheal dilatation balloons, when inflated with an inflator equipped with a pressure manometer, the device generates an outward radial force to dilate the stenotic portion of the airway. The balloon differs from previous devices used for dilatation of tracheal stenosis in that it is modified to have a large central channel when inflated, which allows gas flow through the balloon.

All materials in the device are medical grade and sourced from specialist medical suppliers. The balloons specifically have undergone biocompatibility testing according to ISO 10993-1 (Biological testing of medical devices) and passed all tests. Safety of the devices has been rigorously demonstrated through in vitro bench testing, and balloons have been shown to survive a minimum of 10 inflations to rated burst pressure without bursting. The devices are manufactured by a facility experienced in production of endovascular balloons, in an ISO 14644 Class 7 compliant clean-room in a manufacturing facility that has a certified ISO 13485 quality management system. The balloons are tested as part of an ongoing quality control process, to ensure that tight tolerances are maintained in terms of wall thickness, nominal diameter and rated burst pressure. Furthermore, every tracheal balloon device will have been pressure tested to 16 atm before being used, to ensure that no leaks are present.

The device has been assessed in three previous studies, in manikin, animal and adult human use settings. The studies proved that it is possible to adequately ventilate patients through the modified balloon dilation device. There was no incident of arterial desaturation below 90%. No serious adverse events were recorded.

The study will be conducted over a 12 week period, with an average of 1 patient per week undergoing the procedure at the study site. Recruitment is thus estimated at 12 patients (not procedures).

All research and procedures will take place at Red Cross War Memorial Children's Hospital. Patients will be treated in the operating theatres and will recover in the recovery room, followed by the ENT ward. Patients who have suspected airway narrowing and present to the Department of Otolaryngology will be approached by for potential involvement in the study. The process will be explained obtain written informed consent obtained. The patient will then be treated as per routine care and will be included in the study should inclusion and exclusion criteria be satisfied.

All patients will undergo a thorough routine preoperative assessment. Anaesthesia will be standardized in the absence of specific complication. Routine continuous operative monitoring will be used for all cases, including electrocardiogram, non-invasive automatic blood pressure and pulse oximetry.

A rigid laryngoscope will be inserted into the patient's airway and placed in suspension. The level and severity of the stenosis will be evaluated and the tracheal balloon dilator will be placed at the level of the stenosis under direct vision, using an endoscope. The patient will be kept breathing spontaneously if they do not have a tracheostomy tube. Ventilation will be maintained using a tracheostomy tube, if available.

The balloon will be inflated with water using an inflation device, under direct vision. The pressure in the balloon will be adjusted to 6-8 atmospheres and maintained for at least 1 minute, unless arterial desaturation occurs (SpO2 < 90%) Dilatation will be performed 3 times.

Heart rate and peripheral arterial oxygen saturation will be continuously monitored throughout the procedure. These values will be recorded automatically at one-minute intervals from induction until completion of the dilatation phase, and then at 2.5-minute intervals until recovery from anaesthesia. The stenosis will be graded according to the Myer-Cotton staging system for subglottic stenosis, as well as, the internal diameter of the stenosis being measured (using an endotracheal tube) before and after dilatation.

Adverse events will be recorded in data collection forms. Adverse events will include:

* Arterial desaturation below 90%
* Loss of airway patency
* Inability to ventilate
* Patient coughing or movement
* Haemorrhage
* Inability to pass the bronchoscope
* Balloon failure
* False passage
* Tracheal injury
* Oesophageal injury
* Gastric haemorrhage
* Pneumothorax
* Pneumomediastinum
* Subcutaneous emphysema
* Vocal cord injury
* Mediastinitis
* Chest pain
* Laryngospasm
* Bronchospasm
* Atelectasis
* Pulmonary oedema
* Hypoxia
* Aspiration of water (in case of balloon failure)

Data analysis Data will be collected intraoperatively using a data collection form. This will be transferred to an electronic spreadsheet for analysis. As this is a single-arm study without control devices, no comparative statistics will be calculated. Where appropriate, data will be expressed as mean ± standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Refractory stenosis not amenable to balloon dilatation
* Contraindication to balloon dilatation (long-segment stenosis)
* Patient refusal

Exclusion Criteria:

* Refractory stenosis not amenable to balloon dilatation
* Contraindication to balloon dilatation (long-segment stenosis)
* Patient refusal

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in internal tracheal stenosis diameter | Immediate
  Post-dilation change from pre-dilatation values, measured using Myer-Cotton grade and millimeter value

SECONDARY OUTCOMES:
Peripheral arterial oxygenation | Immediate
  Oxygen saturation nadir as determined by plethysmography
Change in internal tracheal stenosis diameter | 6 weeks post dilatation
  Change from pre- and post-dilatation values, measured using Myer-Cotton grade and millimeter value

CONTACTS AND LOCATIONS:
Overall Officials: Ross Hofmeyr, FCA(SA), Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
The data set will be published after study completion using a medium still to be determined. Data set will be available to other researchers on request.